CLINICAL TRIAL: NCT06781567
Title: A Phase Il Clinical Study to Evaluate the Efficacy and Safety of HG146 Capsules in Participants with Recurrent or Metastatic Adenoid Cystic Carcinoma.
Brief Title: Clinical Trial of HG146 Administered to Participants with Adenoid Cystic Carcinoma
Acronym: HG146
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: HitGen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HG146CN201
Record Dates: First submitted 2025-01-06; First posted 2025-01-17 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-01

CONDITIONS: Adenoid Cystic Carcinoma; Head and Neck Cancer
Keywords: HG146; HG146CN201
MeSH Terms: conditions — Carcinoma, Adenoid Cystic; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clinical Trial of HG146 Administered to participants with Adenoid cystic carcinoma (Experimental): Experimental: HG146 Monotherapy Arm Description: Participants will receive HG146 per os at every two days intervals (qod) for 14 consecutive days,7 days off, 21 days/ cycle.
  Interventions: Drug: HG146

INTERVENTIONS:
Drug: HG146 — HG146 is available as Capsule at a unit dose strength of 5 mg and 10 mg.
  Other Names: HG146 Capsule

SUMMARY:
This is a Phase II, open-label, non-randomized, multicenter study to evaluate the clinical efficacy and safety of HG146 in participants with recurrent or metastatic adenoid cystic carcinoma. This study is divided into two stages. 40 participants will be enrolled in the first stage. The efficacy and safty data will apply to make go or no go decision. Then the second stage will continue to enroll 100 Particapants.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF) and able to comply with study.
* Age ≥18 years, gender unlimited.
* Recurrent or metastatic adenoid cystic carcinoma with evidence of disease progression (imaging progression or clinical evidence of progression) within one year of histological or cytological diagnosis.
* Estimated survival >12 weeks, as determined by the investigator.
* The United States Eastern Cancer Consortium (ECOG) physical status score 0-1.
* Has adequate organ function.
* At least 1 measurable tumor lesion according to RECISTv1.1 criteria.

Exclusion Criteria:

* Symptomatic central nervous system (CNS) metastases that have required steroids within 4 weeks prior to first dose of study treatment.
* Received prior therapies targeting HDAC.
* Chemotherapy was received within 21 days before the first administration of the study treatment, and anti-tumor therapy such as radiotherapy, biotherapy, targeted therapy, and immunotherapy was received within 28 days before the first administration of the study treatment [small molecule targeted drugs, Chinese medicines with anti-tumor indications, and local palliative radiotherapy were 14 times before the first administration of the study drug.
* Used strong CYP3A4 inhibitors or inducers within 7 days before the first use of the investigational drug.
* Major surgery or major injury <=28 days before the first dose of study treatment,or anticipated major surgery during the study.
* Prior allogeneic bone marrow transplantation or other solid organ transplantation
* Active infection requiring systemic treatment.
* Current or past presence of other malignancies (other than adequately treated basal cell or squamous cell carcinoma of the skin and carcinoma in situ of the cervix), unless radical treatment has been performed and there is no evidence of recurrence and metastasis in the last 5 years.
* A person is known to be allergic to any active ingredient or excipient of the investigational drug.
* Pregnant or lactating women.
* patients with drug abuse or chronic alcohol abuse that may affect the evaluation of the test results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | From enrollment to the end of treatment at 4 weeks
  ORR will be assessed by the investigators using RECIST v1.1
6 Months Progression-Free Survival （PFS） | From enrollment to treatment at 6 months.
  PFS will be assessed by the investigators using RECIST v. 1.1

SECONDARY OUTCOMES:
Progression-Free Survival （PFS） | From enrollment to treatment at 12 months
  PFS will be assessed by the investigators using RECIST v1.1
Duration of response (DoR) | From enrollment to the end of treatment at 4 weeks
  DOR will be assessed by the investigators using RECIST v1.1
Disease control rate (DCR) | From enrollment to the end of treatment at 4 weeks
  DCR will be assessed by the investigators using RECIST v1.1
Overall survival (OS) | From enrollment to the end of treatment at 4 weeks
  OS will be assessed by the investigators
Time-to-response (TTR) | From enrollment to the end of treatment at 4 weeks
  TTR will be assessed by the investigators using RECIST v1.1
Population pharmacokinetics (PopPK) | From Cycle1 Day7 to Day13, 21 days per cycle
  PopPK will be detected to predict exposure level of HG146 in human body.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, Principal Investigator — Shanghai Oriental Hospital
Locations (1):
- Shanghai Oriental Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No